CLINICAL TRIAL: NCT02582502
Title: Hyperbaric Oxygen Post Established Stroke - HOPES - Study
Brief Title: Hyperbaric Oxygen Post Established Stroke
Acronym: HOPES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, David Harrison, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H15-00766
Record Dates: First submitted 2015-09-29; First posted 2015-10-21 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Stroke; Ischemic Stroke; Established Stroke
Keywords: Hyperbaric Oxygen; HBOT; Hyperbaric Chamber; Pressurized Oxygen
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): This arm will receive Hyperbaric Oxygen Therapy immediately after consent into study.
  Interventions: Other: Hyperbaric Oxygen
- Wait list Treatment (Other): This arm will receive Hyperbaric Oxygen Therapy two months after consenting into study.
  Interventions: Other: Hyperbaric Oxygen

INTERVENTIONS:
Other: Hyperbaric Oxygen — The only intervention given will be 100% oxygen under hyperbaric pressure.

SUMMARY:
The purpose of this study is to examine the role of Hyperbaric Oxygen Therapy (HBOT) in improving neurological function in patients who are 6 to 36 months post ischemic stroke.

DETAILED DESCRIPTION:
The purpose of this study is to examine the role of Hyperbaric Oxygen Therapy (HBOT) in improving neurological function in patients who are 6 to 36 months post ischemic stroke.

Hyperbaric oxygen therapy (HBOT) involves the administration of inhaled 100% oxygen at increased ambient pressure inside a closed vessel. HBOT produces greatly elevated arterial and tissue oxygen tensions, producing a wide variety of physiological effects at the cellular and sub cellular level. Some of these effects have been postulated to be beneficial in the context of ischemic stroke.

Most of the recovery after stroke occurs in the first 30 to 90 days after the acute event. Recovery is largely based on recovery of brain that is injured, but viable. Physiological imaging studies (PET, EEG) have demonstrated that brain tissue may remain alive but not functional for months or years after ischemic insult.

Subjects will be selected from the stroke population based on an expectation that they would experience a clinically significant improvement. Eligible subjects will have suffered an ischemic stroke involving the cerebral cortex within the last 6 to 36 months. The study will be enrolling 140 subjects and will be randomized to two different treatment arms: experimental group and a waitlist group.

Each subject will receive a series of forty 2 hour treatments, delivered once a day, 5 days a week, within the hyperbaric oxygen chamber.There will be assessments completed before treatment series begins, 3 weeks and 6 weeks into treatment and then again at the end of treatment. After treatment ends, the investigators will conduct these assessments again at 3 months, 6 months, 9 months and 1 year from the date of the participants last treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 19 and 85.
2. Able to speak English and give informed consent or have a substitute decision maker and able to assent.
3. One or more ischemic stroke(s) involving the cerebral cortex or cerebellum within the last 6 to 36 months
4. Able to sit in the chamber with the assistance of a waist and chest strap for 120 minutes.

Exclusion Criteria:

1. Contraindication to HBOT (Appendix C) including:

   1. Untreated collapsed lung (pneumothorax)
   2. Have taken the chemotherapy drug Doxorubicin within 72 hours
   3. Have taken the chemotherapy drug Bleomycin within 4 months
   4. Bowel obstruction
   5. Heart pacemaker of unknown make and model
   6. Pregnancy
   7. Cigarette Smoking
   8. Chronic Obstructive Pulmonary Disease (COPD)
2. Participation in other stroke related studies.
3. Previous history stroke > 36 months prior to study baseline

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2015-10; Primary Completion 2020-01 (Actual); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Change in the Stroke Impact Scale (SIS-16) from baseline over the duration of the study | Pre treatment (Baseline and after waiting period is completed), During Treatment (3 weeks, 6 weeks) and Post Treatment (9 weeks post baseline, 8 months post and 14 months)

SECONDARY OUTCOMES:
National Institute of Health Stroke Scale (NIHSS) | Pre treatment (Baseline and after waiting period) and Post Treatment (9 weeks post baseline, 8 months post and 14 months post)
Nine hole peg board | Pre treatment (Baseline and after waiting period) and Post Treatment (9 weeks post baseline, 8 months post and 14 months post)
Grip Strength | Pre treatment (Baseline and after waiting period) and Post Treatment (9 weeks post baseline, 8 months post and 14 months post)
Berg Balance Test | Pre treatment (Baseline and after waiting period) and Post Treatment (9 weeks post baseline, 8 months post and 14 months post)
6 metre walk test | Pre treatment (Baseline and after waiting period) and Post Treatment (9 weeks post baseline, 8 months post and 14 months post)
6 minutes walk test | Pre treatment (Baseline and after waiting period) and Post Treatment (9 weeks post baseline, 8 months post and 14 months post)
Trail Making Test | Pre treatment (Baseline and after waiting period) and Post Treatment (9 weeks post baseline, 8 months post and 14 months post)
Digital Symbol Substitution Test | Pre treatment (Baseline and after waiting period) and Post Treatment (9 weeks post baseline, 8 months post and 14 months post)
Centre for Epidemiologic Studies Depression Scale (CESD) | Pre treatment (Baseline and after waiting period) and Post Treatment (9 weeks post baseline, 8 months post and 14 months post)
Medical Outcomes Study Short Form (SF-36) | Pre treatment (Baseline and after waiting period) and Post Treatment (9 weeks post baseline, 8 months post and 14 months post)
Montreal Cognitive Assessment (MoCA) | Pre treatment (Baseline and after waiting period) and Post Treatment (9 weeks post baseline, 8 months post and 14 months post)
Health Economics Questionnaire | Pre treatment (Baseline and after waiting period) and Post Treatment (5 months, 8 months, 11 months and 14 months)

CONTACTS AND LOCATIONS:
Overall Officials: David W Harrison, MD,CCFP(EM),FRCPC, Principal Investigator — Vancouver General Hospital and University of British Columbia
Locations (1):
- Vancouver General Hospital - Hyperbaric Unit, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No